CLINICAL TRIAL: NCT01431625
Title: Effects of Exercise Training on Systemic Inflammation an Muscle Repair According to the Chronic Obstructive Pulmonary Disease Phenotype
Brief Title: Effects of Exercise Training on Systemic Inflammation an Muscle Repair According to the Obstructive Chronic Pulmonary Disease (COPD) Phenotype
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Francisco Ortega Ruiz, Head of Section of Pneumology, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/0529
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Obstructive Chronic Pulmonary Disease; Emphysema; Chronic Bronchitis
Keywords: COPD; Exercise Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD with emphysema-predominant (Active Comparator): The degree of involvement of the lung parenchyma and the airway are assessed by computed tomography. The HRCT is performed using 2-mm collimation, scan time 1.0 s, 120 kVp, and 200 mA. Images at three different levels (a cranial section is obtained 1 cm above the superior margin of the aortic arch, a middle section is taken at 1 cm below the carina, and a caudal section is taken approximately 3 cm above the top of the diaphragm) are selected and LAA% is then automatically calculated. The identification threshold of normal lung density and LAA is set at -960 HU. The cut-off level between high or low LAA% is the mean + 2SD of LAA% of the asymptomatic non-COPD smokers.
  Interventions: Other: Combined Training (endurance and strength exercises)
- COPD with airway-predominant (Active Comparator): The degree of involvement of the lung parenchyma and the airway are assessed by computed tomography. The HRCT is performed using 2-mm collimation, scan time 1.0 s, 120 kVp, and 200 mA. Images at three different levels (a cranial section is obtained 1 cm above the superior margin of the aortic arch, a middle section is taken at 1 cm below the carina, and a caudal section is taken approximately 3 cm above the top of the diaphragm) are selected and LAA% is then automatically calculated. The helical scan is performed using 120 kVp, 50 mA, 3-mm collimation, and pith 1.0. The dimensions of the right apical segmental bronchus are measured and WA% is calculated. The cut-off level between high or low WA% is the mean + 2SD of WA% of the asymptomatic non-COPD smokers.
  Interventions: Other: Combined Training (endurance and strength exercises)

INTERVENTIONS:
Other: Combined Training (endurance and strength exercises) — All patients underwent a training program to be held for 12 weeks in sessions of 60 minutes:
  1. .- 20 minutes of bicycle ergometer with an initial load level of about 70% of baseline peak oxygen consumption, increasing the load every two weeks as tolerated.
  2. - Weightlifting in 2 sets of 6 reps of 5 simple exercises. These are held at a station multigimnastyc (CLASSIC Fitness Center, KETTLER) and are as follows: "pulls Chest," "Shoulder press," "Butterfly," "Leg extension" and "Leg curls." The resistance will be increased gradually from 70% of the maximum weight you can lift the patient in a single maneuver (Test 1RM). Every two weeks the maximum weight is re-evaluated to adjust the training load in each patient.
  Other Names: Respiratory Rehabilitation

SUMMARY:
AIM: To identify those mechanisms involved in the systemic and muscular response to exercise treatment, in two different Obstructive Chronic Pulmonary Disease (COPD) phenotypes (emphysema and non-emphysema). The investigators will evaluate the effect of exercise training, on exercise outcomes, peripheral muscle strength measures, dyspnea and quality of life indices, and markers of systemic inflammation and muscle repair.

SUBJECTS: The investigators will study 30 COPD patients in GOLD II-IV stages, with symptomatic disease. Patients will be differentiated into 2 different phenotypes: predominant-emphysema and non-predominant emphysema (15 subjects for each group), according to high resolution computed tomography (HRCT) scanning images, and after the specific analysis with the MeVisPulmo software. After patients are typified, they will be included in the 12- wk training programme. MEASURES(pre&post-training):Basic blood analysis, EKG, spirometry, blood gases, pletysmography, gas diffusion, maximal inspiratory and expiratory pressure (MIP,MEP), bioimpedanciometry, 1RM test and isometric strength determination, 6-min walking test (6MWT), maximal and submaximal cycle-ergometry, and dyspnea using the Mahler's Basal and Transitional Dyspnoea Indexes (BDI/TDI) and quality of life (Chronic Respiratory Disease Questionnaire [(CRDQ]) evaluation. Besides, the investigators will measure blood PCR and cytokines levels (IL6, IL8, IL10, IL12, TNF-α, IGF-1, and MIC-A & MIC-B). Muscle biopsies will be made (quadriceps) for detection of TNF-α, TNFR-I, TNFR-II, IGF-1Ea and MGF, IGF-1R, genes bound to biogenesis, markers of cell lesion-stress and myosin heavy chains (MyHC) type I and II, N-CAM/CD56 and Met & Desmin

DETAILED DESCRIPTION:
STUDY POPULATION: Patients diagnosed COPD using the criteria established by the ATS (American Thoracic Society) and the SEPAR (Spanish Society of Pneumology and Thoracic Surgery) obstruction presenting moderate to severe airway obstruction (FEV1 <60%) and a clinical impact of their disease. Patients should be stable and appropriate therapy, and must not have suffered exacerbations of the disease over a period of three months before the study, and without treatment with oral corticosteroids for at least the same period.

SAMPLE SIZE: 30 patients diagnosed at the Department of Pulmonology, Hospital Virgen del Rocío de Sevilla, informed consent.

Sample size calculation: Analyzing the effect size at the expense of an improvement in the work achieved over 15 W in the stress test, and considering a standard deviation of this parameter + / - 10W, allowing to detect differences in metabolic variables muscle, taking some risks alpha <0.05 and beta < 0, 2 and calculating a percentage of losses of 15%, the investigators estimate a sample size of 15 patients for each group (PC-size).

EXIT CRITERIA OF THE STUDY:

* patient's clinical decompensation
* Loss of 3 or 5 consecutive sessions of the training program discontinued.
* On the initiative of the patient

CHARACTERISTICS OF GROUPS AND STUDY DESIGN:

This is a prospective case-control, with a double oriented ex vivo and in vitro.

Patients differ in COPD "dominance emphysema" (15 patients) or COPD without "predominantly emphysema" (15 patients) achieved according to objective criteria for quantitative methods of a Computed Tomography High Resolution.

The study will follow the recommendations of the Helsinki Declaration on human experimentation and security levels of data protection required by Law 15/1999 of December 13. The study was approved by the ethics committee of our institution and will obtain the informed consent of the individuals recruited.

TRAINING PROGRAM OF THE YEAR:

All patients underwent a training program to be held for 12 weeks in sessions of 60 minutes:

1. .- 20 minutes of bicycle ergometer with an initial load level of about 70% of baseline peak oxygen consumption, increasing the load every two weeks as tolerated.
2. - Weightlifting in 2 sets of 6 reps of 5 simple exercises. These are held at a station multigimnastyc (CLASSIC Fitness Center, KETTLER) and comprise: or simple arm flexion (pull cable to the chest "Chest pulls"): effects on the latissimus dorsa, deltoids and biceps. Sitting facing the tower drive, approaching the bar to the chest and then extending your arms after you return to the starting position.

or simple extension of the arms ("Shoulder press"): Effects on the deltoids and triceps. Sitting upright on the bench and held the weight to shoulder height, there will be extending your arms above your head, slowly returning after bending arms to the starting position.

or arm flexion and extension against resistance (Butterfly "Butterfly"): Effects on the pectoral and deltoid muscles. Sitting upright on the bench with your forearms and elbows on a lever, takes it to the midline, giving way slowly to the starting position.

or leg stretching ("Leg extension"): Effects on the quadriceps. Sitting on the bench leg extension is performed against resistance.

or squats ("Leg curls"): Effects on the biceps femorals and calves. Lying prone on the bench legs are bent against the weight.

The resistance will be increased gradually from 70% of the maximum weight you can lift the patient in a single maneuver (Test 1RM). Every two weeks the maximum weight is re-evaluated to adjust the training load in each patient.

VARIABLES, SAMPLING AND MEASUREMENT:

All patients underwent baseline and after the training program the following tests.

* Analytical elemental, 12-lead electrocardiogram
* Spirometry and bronchodilator test simple: be held in a Datospir 92 at baseline and after administration of 200 micrograms of salbutamol
* Blood gases
* static lung volumes (FRC, RV, TLC) by plethysmography.
* Study of diffusion (DLCO) by single breath technique (equipment Masterlab).
* maximum muscle pressures both inspiratory and expiratory, using a specific gauge (Micro Medical, Rochester, USA) connected to a pressure transducer and a digital recording system.
* chest CT (only at baseline): Phillips Tomoscan with Easy Vision workstation version 4.2 that allows densitometric analysis of lung parenchyma. Quantitative analysis of the degree of emphysema was performed using the software 3D MeVisPULMO (MeVis Research, Research Partner, University of Bremen, Germany). This is a prototype of software that allows functional diagnosis based on CT images and in relation to the anatomical compartments of the lung. Includes automated segmentation of the airway, lungs, lung lobes and segments sublobar approach. This feature makes it especially useful to enhance the diagnostic process in severe lung disease. The analysis software provides a regional assessment MeVisPULMO allows proper parameters measured by CT lung, such as: the total volume, mean density, pixel index or index of bullae (7.22).
* Assessment of muscle strength:

  1. Test one repetition maximum (1 RM test) measures the maximum amount of weight (in kg) that can be raised in a single maneuver using a multigimnastyc station (Classic Fitness Centre, Kettler, Postfach, USA). It can for each of the five exercise of upper and lower limbs that are developed (chest pull, butterfly, shoulder press, leg extension and leg curls).

maximal isometric quadriceps b.strength dominant. There will be a quad chair specially prepared for this procedure (HUR Labs, Sanro) and using a dynamometer cable (Performance recorder). There will be at least 3 maneuvers of maximal isometric force of 5 to 10 sec duration. They are valid exercises that present a variability of less than 10%. The highest value is taken as maximum force.

* Body composition: body compartments estimated greasy, non-fat and body water by bioelectrical impedance power (Bodystat 1500, Isle of Man, United Kingdom). The BMI is calculated by dividing weight (Kg) to height (m2) fat-free mass, Fat Free Mass (FFM) and fat (FM) measured by bioimpedance (). FFM index (FFMi) ratio is calculated by the FFM (kg) and height (m2). The loss of muscle mass is defined as FFM index <16 kg/m2 for men and <15 kg/m2 in women.
* Exercise Test:

  1. Máximal with cycle ergometer and methodology already known (20), including: Determining, from the respiratory gases, oxygen consumption, carbon production and indirect anaerobic threshold, breathing pattern (minute ventilation, tidal volume, frequency breathing), electrocardiographic monitoring and pulse oximetry during exercise with heart rate control, blood pressure and dyspnea Borg scale.
  2. Submáximal of resistance cycle ergometer at 70% load achieved in the ultimate test, with time control of resistance primarily, distance walked and control saturation (pulse oximetry) and heart rate achieved.
  3. Test of the 6-minute walk, according to standard guidelines of the ATS.
* Assessment of dyspnea and quality of life:

  1. Indices of dyspnea and transition rate measures the functional deterioration, the magnitude of the task and the magnitude of effort (Test of Mahler).
  2. Evaluation quality of life based on the specific questionnaire (CRDQ) proposed by Guyatt for COPD patients and modified for your understanding in Spanish-speaking subjects.
* Evaluation of markers of inflammation and catabolism: It will perform a white blood cell count by flow cytometry and measured the levels of CRP in blood samples by quantitative real-time PCR. The detection of various cytokines, IL6, IL8, IL10, IL12, TNF alpha, IGF-1 and MIC-A and MIC-B circulating is carried out by immunosorbent assay (ELISA) using specific kit for each markers.
* Quadriceps Muscle Biopsy: Biopsies were performed in the middle of the thigh, obtaining samples of the vastus lateralis of the quadriceps muscle. Samples were obtained in an outpatient setting. Some of the biopsies were fixed in formalin and included in paraffin blocks and some will freeze with liquid nitrogen and stored at -80 ° C for subsequent use in genetic and immunohistochemical study.

For analysis of expression of genes selected, proceed to extract RNA from tissues previously frozen in liquid nitrogen. This will be used Trizol Reagent (Invitrogen). From isolated RNA was performed reverse transcription using Superscript II RNase kit reverse transcriptase (Invitrogen) and the resulting cDNA was used to carry out real-time quantitative PCR. The PCR reaction was carried out by using fluorochromes such as SYBR Green or Taqman probes (Applied Biosystems). The following will be evaluated based on their genes into the muscle transcriptome:

* TNF-alpha and its two receptors (TNFR-I and TNFR-II), the two isoforms muscle IGF-1 (IGF-1EA and FGM) and its specific receptor (IGF-1R).
* Genes linked to the biogenesis: Paired box gene 7 (Pax7), M-cadherin and Myo-D.
* Markers-cellular stress injury: adult isoforms demiosina heavy chain, both embryonic (MyHC-emb) and perinatal (MyHC-peri).

Immunohistochemical studies were performed in 5 um sections of paraffin tissue blocks previously. These studies will detect markers such as myosin heavy chains (MyHC) I and II (for typing and morphometric study fibrillar) N-CAM/CD 56 and Met (for quantification of satellite cells in muscle tissue) and desmin (for determining the origin muscular). For detection using the standard technique of immunoperoxidase-biotine.avidins (DakoCytomation, Dako Denmark) with antibodies specific for each of the markers.

STATISTICAL ANALYSIS:

For comparison of numeric variables between groups used nonparametric or parametric tests, depending on their distribution (analysis of variance, Student's t test and Mann-Whitney). To analyze the influence of training on the functional and morphometric variables were also conducted an analysis of the percentage change [(post value - value pre / pre value) x 100]. To examine the relationship between different variables using the Pearson correlation coefficients or Spearman, according to the distribution thereof. There will also be a multivariate analysis, multiple regression. Be considered statistically significant at p <0.05. The dispersion of a mean value is expressed as mean ± standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients diagnosed according to criteria established by the ATS (American Thoracic Society) and the SEPAR (Spanish Society of Pneumology and Thoracic Surgery) obstruction presenting moderate to severe airway obstruction (FEV1 <60%) and a clinical impact of their disease. Patients should be stable and appropriate therapy, and must not have suffered exacerbations of the disease over a period of three months before the study, and without treatment with oral corticosteroids for at least the same period.

Exclusion Criteria:

* Other cardio-respiratory diseases, cardiovascular, neuromuscular or metabolic might interfere with the results.
* Systemic diseases, alcohol intake (> 80 g / day) or treatment with drugs with potential effect on muscle structure
* Inability or disagree to participate in an exercise program.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in TNF-alpha and its receptors, muscle isoforms of IGF-1 and its receptor in samples of quadriceps muscle satellite cells at 3 moths. | Baseline and end of follow-up period of 3 moths
  Compare these values according to the phenotype of the patient (airway-predominant vs. emphysema-predominant) and assess the effect of the training program, according to the phenotype, the regenerative potential and muscle remodeling.

SECONDARY OUTCOMES:
Pax7, M-cadherin and Myo-D and its receptor in samples (molecules and repair-myogenesis) of quadriceps muscle satellite cells. | Baseline and end of follow-up period of 3 moths
  Compare these values according to the phenotype of the patient (airway-predominant vs. emphysema-predominant) and assess the effect of the training program, according to the phenotype, the regenerative potential and muscle remodeling.
MIC-A and MIC-B soluble in serum. | Baseline and end of follow-up period of 3 moths.
  Compare these values according to the phenotype of the patient (airway-predominant vs. emphysema-predominant) and assess the effect of the training program, according to the phenotype. Determine whether the presence of these substances impact in terms of exercise capacity, nutritional status and muscle function.
CRP, IL6, IL8, IL10, IL12, TNF alpha, IGF-1 (systemic inflammatory profile) in serum. | Baseline and end of follow-up period of 3 moths.
  Compare these values according to the phenotype of the patient (airway-predominant vs. emphysema-predominant) and assess the effect of the training program, according to the phenotype. Determine whether the presence of these substances impact in terms of exercise capacity, nutritional status and muscle function.

CONTACTS AND LOCATIONS:
Overall Officials: Ortega F Ruiz, Doctor, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Sevilla, Spain